CLINICAL TRIAL: NCT05596188
Title: Status and Independent Risk Factors of Preoperative Anxiety in Adults Undergoing Non-cardiac Surgery: a Cross-sectional Study
Brief Title: Anxiety Before Non-cardiac Surgery in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SSY04070224
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Myoma of Uterus; Colon Cancer; Gastric Carcinoma; Prostate Cancer; Femoral Head Necrosis
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adult patients undergoing elective non-cardiac surgery were enrolled. Anxiety before the operation was evaluated by The State Anxiety Inventory (S-AI). Logistics regression would be used for identifying the independent factors of preoperative anxiety and prediction model would be established.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing elective with general anesthesia surgery (gynecologic oncology, general surgery, orthopedics and urinary);
2. The estimated operation time is more than 2 hours. 3)18≤ age ≤ 80;

4)be able to communicate normally in daily life, without serious hearing and visual impairment; 5)ASA:I-II; 6)sign informed consent and volunteer to participate in this study.

Exclusion Criteria:

1. Having a history of brain diseases, such as stroke, epilepsy, psychosis other history of neuropsychiatry.
2. Patients with serious diseases of heart, liver, lung, kidney or other organs.
3. Having a definite diagnosis of cognitive impairment, such as Alzheimer's disease;
4. Those who use sedatives before evaluation in this study;
5. Drug addicts;
6. Alcoholics;
7. pregnant women;
8. participated in other clinical trials as a subject in the past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who met the eligibilty criteria for elective surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-10-17 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Independent risk factors of preoperative anxiety and establishment of prediction model | From the 1 day before surgery to 7 days after surgery or discharge, whichever came first
  To identify the independent factors related to preoperative anxiety, which would be analyzed by Logistic regression according to anxiety or not before surgery evaluated by the State anxiety inventory（20-80，lower is better) . Meanwhile, the prediction model of preoperative anxiety would be established based on independent factors.

SECONDARY OUTCOMES:
Incidence of preoperative anxiety | The 1 day before surgery
  The State anxiety inventory (20-80，lower is better) was used to investigate the incidence of Preoperative anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China